CLINICAL TRIAL: NCT06162182
Title: Comparative Evaluation of an Electrical Impedance Device Versus Digital Radiography in Estimation of Remaining Dentin Thickness in Carious Posterior Permanent Teeth (Diagnostic Accuracy Trial)
Brief Title: Comparative Evaluation of an Electrical Impedance Device Versus Digital Radiography in Estimation of Remaining Dentin Thickness
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rawda Hesham Abd ElAziz (Other)
Responsible Party: Sponsor-Investigator, Rawda Hesham Abd ElAziz, Lecturer, Conservative dentistry department, Faculty of Dentistry, Cairo University., Cairo University
Organization: Cairo University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: CEBD 4/2023
Record Dates: First submitted 2023-11-14; First posted 2023-12-08 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Caries,Dental; Deep Caries
Keywords: electrical impedance device (prepometer); digital radiography; remaining dentin thickness
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The assessors will not be blind about the type of intervention/control assessment methods due to different application methods. However it will not be allowed amongst the examiners to exchange any information throughout the entire study period
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reference test: Radiographic examination (Experimental)
  Interventions: Diagnostic Test: Reference test: Digital Radiographic examination
- Index test: electrical impedance device, Prepometer (Experimental)
  Interventions: Diagnostic Test: electrical impedance device,

INTERVENTIONS:
Diagnostic Test: electrical impedance device, — The electrical resistance of the residual dentine underneath each measurement point was determined between an electrode and the crown pulp (Prepometer, Hager & Werken, Duisburg, Germany). Assigning the electrical resistance of the dentin. high values are considered to represent more residual dentine than low values.
  Other Names: Prepometer
  Arms: Index test: electrical impedance device, Prepometer
Diagnostic Test: Reference test: Digital Radiographic examination — A digital periapical radiograph using paralleling technique was taken
  Arms: Reference test: Radiographic examination

SUMMARY:
The research question was that in patients with carious posterior permanent teeth, would the electrical impedance device be as valid as digital radiography in estimation of remaining dentin thickness? The proposed hypothesis was null.

ELIGIBILITY:
Inclusion Criteria:

* Participants eligible for this study were those aged from 18 y to 28 y,
* willing to join the study
* with clinically detectable occlusal or proximal carious vital permanent molar teeth with closed apex and healthy periodontal supporting.
* The minimum extension of the carious cavity should be at least 1 mm in width to accommodate with the probe of the prepometer

Exclusion Criteria:

* Excluded participants were those with poor oral hygiene,
* severe medical complications,
* showing signs and symptoms of irreversible or necrotic pulp pathology also when the affected tooth was with extended buccal or lingual caries, extending clinically beyond ¼ dentin thickness or previously restored.

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 67 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-12-20 (Estimated)

PRIMARY OUTCOMES:
validity of the two devices | Through study completion, an average of 1 year
  Level of agreement between the digital radiograph and the device in measurement of remaining dentin thickness

SECONDARY OUTCOMES:
Patients satisfaction between two devices | Through study completion, an average of 1 year
  By visual analogue scale Visual Analog Scale (VAS) which is a 100 mm straight horizontal line with the left end indicating •not at all satisfied- and the right end "very satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Rawda Hesham Abd ElAziz, PhD, Principal Investigator — Lecturer, Conservative dentistry department, Faculty of Dentistry, Cairo University.
Locations (2):
- Egypt (2):
  - Faculty of Dentistry, Cairo
  - Cairo University, Cairo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Krause F, Braun A, Eberhard J, Jepsen S. Laser fluorescence measurements compared to electrical resistance of residual dentine in excavated cavities in vivo. Caries Res. 2007;41(2):135-40. doi: 10.1159/000098047. PMID 17284915